CLINICAL TRIAL: NCT02539784
Title: Thoracic Spinal Cord Stimulation as a Symptomatic Treatment for Advanced Parkinson's Disease: A Phase I Safety and Efficacy Study
Brief Title: Thoracic Spinal Cord Stimulation as a Symptomatic Treatment for Advanced Parkinson's Disease
Acronym: SpinalPark
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P121205
Record Dates: First submitted 2015-07-27; First posted 2015-09-03 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson
Keywords: stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Cord Stimulation (Experimental)
  Interventions: Device: Kit for Spinal Cord Stimulator System " SCS Systems " : PRECISION® System

INTERVENTIONS:
Device: Kit for Spinal Cord Stimulator System " SCS Systems " : PRECISION® System — 3 frequencies of SCS are tested for each patient : 50, 100 and 130 Hz
  Other Names: Boston Scientific Device

SUMMARY:
Following the so call "honey moon" period, motor symptoms of Parkinson's Disease (PD) become difficult to control with dopaminergic treatments alone. Deep brain stimulation (DBS) of the subthalamic nucleus and internal globus pallidus helps to treat fluctuating parkinsonian patients restoring a decent quality of life. However, DBS need a long, complex and invasive surgery to succeed. Thus, there is a critical need to develop alternative treatments, more accessible and less invasive. Thoracic posterior spinal cord stimulation has been used for decades to treat chronic neuropathic pains. Safety and efficacy have already been demonstrated in neuropathic pain. Experimentally, SCS has also demonstrated to improve locomotor activity in two different rodents' models of parkinson's disease. The purpose of this study is to determine whether thoracic SCS is safe and could induce a benefit motor parkinsonian symptoms without any impact on cognitive function and axial disability.

DETAILED DESCRIPTION:
The present pilot study will enroll 6 patients suffering from advanced Parkinson Disease (PD). Investigator will assess the safety, tolerance and efficacy of Spinal Cord Stimulation (SCS) with frequencies of 50, 100 and 130 Hz in a shuffle randomized for each patient. Briefly, each frequency will be evaluated immediately after and 4 weeks following SCS initiation with UPDRS-III, pain scales, and Hauser's diary. The best frequency for each patient will be then selected and maintained activated for 12 additional weeks. At the end of these 12 weeks, new assessment including UPDRS, visual pain scale, "SAINT-ANTOINE" Pain Questionary, PDQ-39 (quality of life), daily L-dopa equivalent dose, MDRS (cognitive status), LARS (apathy status) and MADRS (depression status) will be compared to the inclusion data of each patient. Primary endpoints include the safety of thoracic SCS by collected the number of adverse event and the efficacy by measuring the UPDRS-III OFF med/ON stim at 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 45 to 69 years old
* Affiliated to the French social health care system
* Menopausal or under contraception for women
* Parkinson's disease according to UK PDSBB's criteria with diagnosis for ≥ 5 years
* OFF UPDRS-III ≥ 25
* Acute dopa-response ≥ 50% for UPDRS-III in an L-Dopa challenge
* Fluctuations with periods off ≥ 25% of the time of awakening or dyskinesia ≥ 25%
* 3≤ Hoehn & Yahr ≤ 4
* No change in anti-parkinsonian drugs in the last month
* Informed consent signed for the study

Exclusion Criteria:

* Patients major protected
* Pregnancy
* Deep brain stimulation or other neurosurgical treatment
* MDRS Score < 130 or depression scale MADRS ≥ 20
* Respiratory insufficiency (surgery belly decubitus)
* Abnormalities on brain MRI which evoke a secondary parkinsonian syndrome
* Spinal cord's injury on MRI or posterior cordonal's pathology on sensitive evoked potential
* Neuropathy on EMG
* Prior spinal surgery and spinal pathology at the dorsal level
* Patients having already been included in therapeutic studies
* Patient with a cardiac pacemaker, a defibrillator or any other implanted active pacemaker
* Patient requiring diathermy process
* Patient having a pathology requiring an MRI follow-up care

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of severe adverse events and adverse events reported | at week 30

SECONDARY OUTCOMES:
Tolerance and global statement | After surgery (DO), at week 4, 8, 13, 18 and 30
  Clinical assessment
Difference of UPDRS-III scores with and without stimulation in ON or OFF medication state | At W4, W9, W14,W30
Difference of UPDRS-III scores without stimulation and after 4 weeks of continuous stimulation in ON or OFF medication state | At W4, W8, W9, W13, W14,W18
Difference of global UPDRS between screening and others visits, in OFF and ON medication state | At W-4, W8, W13, W18,W30
Difference of Walking Time Measurement scores with and without stimulation in ON or OFF medication state | At W4, W9, W14,W30
Difference of Walking Time Measurement scores without stimulation and after 4 weeks of continuous stimulation in ON or OFF medication state | At W4, W8, W9, W13, W14,W18
Pain assessment using visual pain scale and Saint Antoine Pain Questionnaire | After 4, 9, 13 and 30 weeks after surgery
Paresthesia assessment using visual pain scale and Saint Antoine Pain Questionnaire | After 4, 9, 13 and 30 weeks after surgery
Clinical abnormalities demonstrated during a comprehensive sensitive examination | At W4, W8, W13, W18, W30
Differences of MDRS, LARS, MADRS, PDQ-39 scores between screening and the end of the study | At W-4 and W30
Change of daily L-Dopa equivalent dose | At W4, W8, W13, W18, W30

CONTACTS AND LOCATIONS:
Overall Officials: Claire Thiriez, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France